CLINICAL TRIAL: NCT05067556
Title: Creating a Pathway for Disease-Free Cancer Survivors to Decrease Long-term Opioid Use
Brief Title: Decreasing Long-term Opioid Use in Cancer Survivors
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staffing
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MCC-21-18366
Record Dates: First submitted 2021-09-16; First posted 2021-10-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Pain; Chronic Pain; Cancer Pain; Survivorship
Keywords: Commitment Therapy
MeSH Terms: conditions — Pain; Chronic Pain; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Acceptance and Commitment Therapy for Chronic Pain (ACT-CP)
  Interventions: Behavioral: Acceptance and Commitment Therapy for chronic pain (ACT-CP)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for chronic pain (ACT-CP) — Delivered virtually via Zoom or via telephone on an individual level; 30-minute sessions led by a trained psychologist and occur weekly for 6 weeks.

SUMMARY:
This is a feasibility pilot trial assessing a behavioral intervention for chronic pain among disease-free cancer survivors to decrease long-term opioid dependence.

DETAILED DESCRIPTION:
To assess the feasibility and acceptability of implementing brief Acceptance and Commitment Therapy for chronic pain (ACT-CP) in a Survivorship clinic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer of any type, currently in remission, having completed active primary therapy. Patients on oral adjuvant hormone therapy will still be eligible.
* Completed active therapy must have been curative in intent (for example stage IV cancer patients such as head and neck cancer patients treated with curative intent are eligible).
* Self-reported cancer pain for >= 3 months
* Opioid use >= 5MME/day (morphine milligram equivalents) as prescribed by physician for cancer-related pain for at least 6 months beyond completion of their cancer treatment
* VCUHealth system patient

Exclusion Criteria:

* History of opioid use prior to cancer diagnosis
* Anyone with prior history of substance use disorder or currently enrolled in a methadone program
* Anyone with schizophrenia or bipolar disorder
* Current utilization of psychotherapy services for pain, depression, anxiety, and/or PTSD
* Cognitive concerns that would prevent meaningful engagement in treatment
* Inability to converse in English
* Lack of working telephone and Internet connection (must have at least one or the other)
* Anyone found to have progression of cancer
* Anyone diagnosed with cancer recurrence or new cancer during their study period
* Documented diagnosis of or positive screen for current substance use disorder (score >5 on the Drug Abuse Screening Test-10 [DAST-10])
* Anyone scoring >=8 on ORT indicating very high risk for opioid abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment yield of participants contacted | 12 Months
  Study feasibility will be assessed by tracking the number of patients contacted
Recruitment yield of participants consented | 12 Months
  Study feasibility will be assessed by tracking the number of participants that consent to enroll in the trial.
Recruitment yield number of participants enrolled | 12 Months
  Study feasibility will be assessed by recruitment yield, i.e., tracking the number of participants who initiated treatment.
Session Attendance | 6 Weeks
  Study feasibility will be assessed by tracking the number of participants attend each intervention session over the course of the 6-week intervention period.
Participant Satisfaction | 6 Weeks
  Study acceptability will be assessed by administering a post-intervention satisfaction survey which asks about satisfaction with the program including perceived efficacy and suggestions for improvement.

SECONDARY OUTCOMES:
Pain Intensity | 6 Weeks
  Preliminary efficacy of acceptance and commitment therapy for chronic pain (ACT-CP) will be assessed by analyzing change in self-reported pain scores using The Patient-Reported Outcome Measurement Information System short form 3a v1.0 (PROMIS). This tool measures how much a person hurts.
Opioid Use Frequency | 6 Weeks
  Preliminary efficacy of acceptance and commitment therapy for chronic pain (ACT-CP) will be assessed by self-reported opioid use frequency weekly throughout the intervention period.
Pain interference | 6 Weeks
  Preliminary efficacy of acceptance and commitment therapy for chronic pain (ACT-CP) will be assessed by analyzing pain interference using the PROMIS short form 8a. The PROMIS Pain Interference instrument measures the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities.
Opioid Refill Frequency | 6 Weeks
  Frequency of opioid refills will be assessed via pharmacy records available in patients' EMR

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hong, MD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data at this time